CLINICAL TRIAL: NCT06674395
Title: Cross Cultural Validation of Urdu Version of Leicester Cough Questionnaire (LCQ)
Brief Title: Validation of Urdu Version of Leicester Cough Questionnaire (LCQ)
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/24/0316
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: COPD
Keywords: cough; patient reported outcome measures; pulmonary diseases; validation study; translations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Leicester Cough Questionnaire (LCQ) is a patient reported, 19-item tool, and it comprised physical, psychological, and social elements. The objective of the study is to cross culturally adapt LCQ in Urdu language and to find the reliability and validity in patients of COPD.

It is a three-stage study. Leicester Cough Questionnaire (LCQ) will be adapted in Urdu and will be first tested for its content validity by using content validity index (CVI).

In the second stage, the Urdu version of the Leicester Cough Questionnaire (LCQ) will be pilot run; tested for its validity and reliability. In the third stage, the Urdu version of the Leicester Cough Questionnaire (LCQ) will be tested for its validity and reliability in patients with COPD.

114 Patients with COPD will be selected according to inclusion criteria. Intra class correlation coefficient (ICC), Cronbach's alpha and factor analysis will be used to analyze the data.

DETAILED DESCRIPTION:
Cough is a common symptom of asthma, COPD, and bronchiectasis, little is known about how it affects health status; therefore any negative effects may go unnoticed in these situations. Leicester Cough Questionnaire (LCQ) is a patient reported, 19-item tool, and it comprised physical, psychological, and social elements. To the extent of author's knowledge, this widely used Leicester Cough Questionnaire (LCQ) has not been translated and validated for Urdu-speaking patients with COPD.

The objective of the study is to cross culturally adapt LCQ in Urdu language using international guidelines used for translation of instrument from its source language to target language and to find the reliability, validity, sensitivity, and specificity of the Urdu version of Leicester Cough Questionnaire (LCQ) in patients of COPD. It is a three-stage study.

Leicester Cough Questionnaire (LCQ) will be adapted in Urdu and will be first tested for its content validity by using content validity index (CVI). In the second stage, the Urdu version of the Leicester Cough Questionnaire (LCQ) will be pilot run; tested for its validity and reliability. In the third stage, the Urdu version of the Leicester Cough Questionnaire (LCQ) will be tested for its validity and reliability in patients with COPD. 114 Patients with COPD will be selected according to inclusion criteria. Intra class correlation coefficient (ICC), Cronbach's alpha and factor analysis will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with GOLD II, III and IV Chronic Obstructive Pulmonary Diseases
* Having age18 years or more
* subjects having chronic cough (> 8 weeks)
* Subjects understanding Urdu

Exclusion Criteria:

* A previous history of other lung disorders
* Pregnant females, subjects having Infections
* Any systemic disorder which is unstable
* Subjects who are not willing to participate
* subject with Cognitive & speech disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Chronic Obstructive Pulmonary Diseases
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Leicester Cough Questionnaire (LCQ) | At Baseline and after 1 week
  LCQ is a 19-item cough measuring tool, created in 2003 by Birring et al., and it comprised physical, psychological, and social elements.
St. George Respiratory Questionnaire | At Baseline and after 1 week
  Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Zia, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Gujranwala Medical College Teaching Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polley L, Yaman N, Heaney L, Cardwell C, Murtagh E, Ramsey J, MacMahon J, Costello RW, McGarvey L. Impact of cough across different chronic respiratory diseases: comparison of two cough-specific health-related quality of life questionnaires. Chest. 2008 Aug;134(2):295-302. doi: 10.1378/chest.07-0141. Epub 2007 Dec 10. PMID 18071022
- [Background] Young EC, Smith JA. Quality of life in patients with chronic cough. Ther Adv Respir Dis. 2010 Feb;4(1):49-55. doi: 10.1177/1753465809358249. Epub 2010 Jan 5. PMID 20051447
- [Background] Wang Z, Wang M, Wen S, Yu L, Xu X. Types and applications of cough-related questionnaires. J Thorac Dis. 2019 Oct;11(10):4379-4388. doi: 10.21037/jtd.2019.09.62. PMID 31737324
- [Background] Birring SS, Prudon B, Carr AJ, Singh SJ, Morgan MD, Pavord ID. Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax. 2003 Apr;58(4):339-43. doi: 10.1136/thorax.58.4.339. PMID 12668799
- [Background] Huisman AN, Wu MZ, Uil SM, van den Berg JW. Reliability and validity of a Dutch version of the Leicester Cough Questionnaire. Cough. 2007 Feb 21;3:3. doi: 10.1186/1745-9974-3-3. PMID 17313670
- [Background] Gao YH, Guan WJ, Xu G, Gao Y, Lin ZY, Tang Y, Lin ZM, Li HM, Luo Q, Zhong NS, Birring SS, Chen RC. Validation of the Mandarin Chinese version of the Leicester Cough Questionnaire in bronchiectasis. Int J Tuberc Lung Dis. 2014 Dec;18(12):1431-7. doi: 10.5588/ijtld.14.0195. PMID 25517807
- [Background] Sonnerfors P, Faager G, Einarsson U. Translation of the Leicester Cough Questionnaire into Swedish, and validity and reliability in chronic obstructive pulmonary disease. Disabil Rehabil. 2018 Nov;40(22):2662-2670. doi: 10.1080/09638288.2017.1353648. Epub 2017 Jul 20. PMID 28728439
- [Background] Dabrowska M, Krakowiak K, Radlinska O, Rybka A, Grabczak EM, Maskey-Warzechowska M, Korczynski P, Birring SS, Krenke R. Validation of the Polish Version of the Chronic Cough Quality of Life Questionnaire (Leicester Cough Questionnaire). Adv Clin Exp Med. 2016 Jul-Aug;25(4):649-53. doi: 10.17219/acem/59512. PMID 27629838
- [Background] Kwon JW, Moon JY, Kim SH, Song WJ, Kim MH, Kang MG, Lim KH, Lee SH, Lee SM, Lee JY, Kwon HS, Kim KM, Kim SH, Kim SH, Jeong JW, Kim CW, Cho SH, Lee BJ; Work Group for Chronic Cough, the Korean Academy of Asthma, Allergy and Clinical Immunology. Reliability and validity of a korean version of the leicester cough questionnaire. Allergy Asthma Immunol Res. 2015 May;7(3):230-3. doi: 10.4168/aair.2015.7.3.230. Epub 2014 Dec 18. PMID 25749761
- [Background] Reychler G, Schinckus M, Fremault A, Liistro G, Pieters T. Validation of the French version of the Leicester Cough Questionnaire in chronic obstructive pulmonary disease. Chron Respir Dis. 2015 Nov;12(4):313-9. doi: 10.1177/1479972315602618. Epub 2015 Sep 7. PMID 26346891